CLINICAL TRIAL: NCT04120142
Title: Effect of Inspiratory Muscle Training During PR on Dyspnoea and Exercise Tolerance in Chronic Obstructive (COPD)
Brief Title: Effect of Inspiratory Muscle Training During PR on Dyspnoea and Exercise Tolerance in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Bilel Tounsi, PhD, Faculty of Medicine, Sousse
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: COPD-DYS
Record Dates: First submitted 2019-09-30; First posted 2019-10-09 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; IMT; 6MWT; Dyspoea; SGRQ
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMT goup (Experimental): Inspiratory muscle training + aerobic exercice
  Interventions: Other: Pulmonary rehabilitation+IMT
- Control group (Active Comparator): aerobic exercice
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation+IMT — The experimental group receives inspiratory muscle training and aerobic exercise.
  Arms: IMT goup
Other: Pulmonary rehabilitation — The Active Comparator group received only aerobic exercise.
  Arms: Control group

SUMMARY:
Chronic obstructive pulmonary disease is a respiratory disease that results in progressive airflow limitation and respiratory distress.

The benefit of inspiratory muscle training (IMT) combined with a pulmonary rehabilitation programme is uncertain. The investigators aimed to demonstrate that, in patients with obstructive pulmonary disease, IMT performed during a PRP is associated with an improvement of dyspnoea and exercise tolerance.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of the inspiratory muscle training (with incremental load every two weeks in two months) performed during pulmonary rehabilitation on dyspnoea, 6 minutes walk test and quality of life using the St George's respiratory questionnaire (SGRQ) in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Were COPD diagnosed by pulmonary function testing
* Clinically stable
* Abscence of other obstructive diseases
* Signed written consert

Exclusion Criteria:

* Were previous pneumonectomy or lobectomy in the past 6 months
* spontaneous risk of pneumothorax or rib fracture
* Incapacity to follow a standard rehabilitation programme (locomotor deficits, acute cardiac failure and acute exacerbation of COPD at the beginning of the programme)
* The absence of written informed consent.

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Dyspnoea | Baseline, After 2 months
  The dyspnoea were measured before and after the 6 minutes walk test
Inspiratory muscle strength | Baseline, After 2 months
  The inspiratory muscle strength were measured by maximal inspiratory pressure test

CONTACTS AND LOCATIONS:
Locations (1):
- Bilel TOUNSI, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langer D, Charususin N, Jacome C, Hoffman M, McConnell A, Decramer M, Gosselink R. Efficacy of a Novel Method for Inspiratory Muscle Training in People With Chronic Obstructive Pulmonary Disease. Phys Ther. 2015 Sep;95(9):1264-73. doi: 10.2522/ptj.20140245. Epub 2015 Apr 9. PMID 25858974
- [Background] Beaumont M, Mialon P, Le Ber C, Le Mevel P, Peran L, Meurisse O, Morelot-Panzini C, Dion A, Couturaud F. Effects of inspiratory muscle training on dyspnoea in severe COPD patients during pulmonary rehabilitation: controlled randomised trial. Eur Respir J. 2018 Jan 25;51(1):1701107. doi: 10.1183/13993003.01107-2017. Print 2018 Jan. PMID 29371379
- [Background] Ambrosino N. Inspiratory muscle training in stable COPD patients: enough is enough? Eur Respir J. 2018 Jan 25;51(1):1702285. doi: 10.1183/13993003.02285-2017. Print 2018 Jan. No abstract available. PMID 29371389